CLINICAL TRIAL: NCT04303871
Title: Comparison Between Invasive and Non-invasive Assessment of Blood Pressure in Hypertensive Disorders of Pregnancy
Brief Title: Invasive Versus Non-invasive Assessment of Blood Pressure in Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Khairy Mohamed Hassan, assistant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17101032
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Hypertension in Pregnancy
Keywords: invasive blood pressure; non-invasive blood pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Active Comparator): pregnant female with hypertension admitted in ICUfor control of BP invasive assessment of BP by radial cannulation was compared against non-invasive assessment of BP by an automated oscillometric BP device (Mobil-O-Graph )
  Interventions: Diagnostic Test: Invasive blood pressure assessment by radial artery canulation
- control (Placebo Comparator): matched control females of the same age but not pregnant invasive compared to non-invasive measurement of BP by same technique
  Interventions: Diagnostic Test: Invasive blood pressure assessment by radial artery canulation

INTERVENTIONS:
Diagnostic Test: Invasive blood pressure assessment by radial artery canulation — radial artery canula used to measure central blood pressure compared to non invasive automated device to measure BP in pregnant females
  Other Names: non invasive assement of BP by automated ossilometric M-Moblie graph

SUMMARY:
Hypertensive disorders of pregnancy are important causes of maternal morbidity and mortality worldwide. Hypertension is one of the most commonly reported health conditions among pregnant women and complicates 5-10% of all pregnancies.(Martin et al., 2009) (Wagner et al., 2007) The measurement of central BP in hypertensive patients became more important because of its predictive value for cardiovascular events. Direct intra-arterial readings are considered to be the gold standard method for blood pressure measurement but because arterial cannulation is associated with risks, alternative non-invasive blood pressure measurements may be used. (Araghi et al., 2006) In our study, the investigator aimed to assess the accuracy of non-invasive central blood pressure by oscillometric automated device (Mobil O graph) in comparison to the invasive blood pressure measurement by arterial cannulation in patients with hypertensive disorders in pregnancy.

the investigators enrolled 100 pregnant women and 10 healthy non-pregnant women as a control group, central blood pressure was measured invasively by arterial cannula and non-invasively by oscillometric automated device (Mobil O Graph).

the investigatorshave found a high correlation between non-invasive central blood pressure measurements and invasively measured both systolic (r 0.968, p=0.000) and diastolic (r 0.687, p=0.000).

DETAILED DESCRIPTION:
Study Methods:

All patients included in our study were subjected to the following:

1. Full history taking including:

   Age, full obstetric history including (number of previous pregnancies and abortions), history of previous illness, duration of pregnancy.

   Risk factors for developing hypertension as Diabetes Mellitus (DM), history of chronic hypertension, anti-hypertensive treatment, history of HTN during previous pregnancies.
2. Full physical examination:

   On admission: Patient's weight and height were obtained to calculate Body surface area (BSA) Vital signs assessment regarding arterial pulse, arterial blood pressure measurement using mercury sphygmomanometer and proper arm cuff according to the recent guidelines of arterial hypertension General and local cardiac examination.
3. Investigations : the followings were done at time of hospital admission:

   1. Urine analysis: was done to all participants to exclude the presence of albuminuria
   2. Echocardiography:

All participants underwent resting transthoracic 2D echocardiography, Scans were acquired by a standard parasternal/apical views using (VIVID S5 instrument, GE Medical Systems, Horten, Norway) with subjects in the left lateral decubitus position.

4) Blood pressure assessment: was done after control of blood pressure by different anti-hypertensive drugs mostly on 3rd- 4th day of admission.

1. Office blood pressure measurement: BP in pregnancy was measured in the sitting position (or the left lateral recumbent during labour) with an appropriately sized arm cuff at heart level and using Korotkoff V for DBP. Manual auscultation was the only method used as it remains the gold standard for BP measurement in pregnancy, because automated devices tend to under-record the BP and are unreliable in severe preeclampsia.
2. Non-invasive central BP monitoring: measured by MOBIL-O-GRAPH:

   * The non-invasive assessment of estimated PWV was performed in a quiet, temperature-controlled examination room
   * Three measurements were taken with a 2-min break between them. The procedure was performed with the patient in a sitting position and using an adequately sized cuff. The Mobil-O-Graph 24h NG (IEM, Stolberg, Germany) with inbuilt ARCSolver (Austrian Institute of Technology, Vienna, Austria) This device is a commercially available brachial oscillometric blood pressure monitor with Food and Drug Administration and Conformite´ Europe´enne approval. Its blood pressure detection unit is validated according to the British Hypertension Society and European Society of Hypertension recommendations. Algorithms were used to obtain conventional blood pressure readings such as brachial systolic and diastolic pressures. In the second step, the brachial cuff is inflated to the diastolic blood pressure level and held for about 10s to record the pulse waves. Subsequently, central pressure curves obtained through a transfer function from the peripheral reading are plotted. To estimate aPWV, the ARCSolver method utilizes several parameters from pulse wave analysis and wave separation analysis combined in a proprietary mathematical model, whereby the major determinants are age (Mendes, 2015) , central pressure, and aortic characteristic impedance.
3. Invasive blood pressure measurement:

Cannulation technique:

Percutaneous cannulation is performed under aseptic conditions, using the radial artery. The hand and forearm are affixed to an arm board, with the wrist dorsiflexed over a bandage roll. The thumb should be immobilized as well, to ensure proper anchorage of the artery. the investigators infiltrate subcutaneously with 2% lidocaine as a local anaesthetic, it helps also to minimize arterial spasm.

Using palpation of the artery as a guide, the cannula (20-gauge Teflon cannula) is advanced at a 20° angle to the skin until the arterial wall is pierced. The stylet is then held fixed and the cannula advanced up the arterial lumen.

The cannula was connected to a disposable tubing system and flushed intermittently with heparinized 0.9% saline solution. This helped prevent occlusion of the cannula by thrombus .The tubing should be stiff and not contain any bubbles in order to minimize resonance and damping.

The liquid within the tubing was connected to a transducer (Auto Transducer®; ACE Medical, Inc., Goyang, Korea). The transducer needs to be kept horizontally level with the patient; traditionally, the right atrium because raising or lowering the transducer relative to the patient will alter the reading. Zeroing was performed by opening the transducer to atmospheric pressure and electronically zeroing the system.

The arterial blood pressure signals were recorded and displayed on a bedside monitor (GE Datex-Ohmeda S/5TM Anaesthesia Monitor, Helsinki, Finland).The whole tubing system was flushed with sterile normal saline to eliminate air bubbles and tested for system loss.

ELIGIBILITY:
Inclusion Criteria:

All Pregnant women diagnosed to have hypertensive disorders of pregnancy (chronic HTN, gestational HTN, pre-eclampsia or eclampsia) after control of hypertension using anti-hypertensive drugs.

Exclusion Criteria:

* Patients with previous cardiac diseases.
* Chronic kidney disease (CKD) which is defined as kidney damage or glomerular filtration rate (GFR) <60 mL/min/1.73 m2 for 3 months or more, irrespective of cause.
* Any disease requiring the use of anti-inflammatory medication, any other endocrine disease such as hyperthyroidism.
* Conditions that prevent invasive blood pressure measurement (arterial cannulation) as severe bleeding disorders.
* Patients refusing to join the study.
* Any associated severe comorbidities have been excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only females included during pregnancy
Enrollment: 117 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
assess accuracy of non-invasive central blood pressure | 12 months
  to assess accuracy of non-invasive central blood pressure by oscillometric automated device (Mobil O graph) in comparison to the invasive blood pressure measurement by arterial cannulation in patients with hypertensive disorders in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] KROEKER EJ, WOOD EH. Comparison of simultaneously recorded central and peripheral arterial pressure pulses during rest, exercise and tilted position in man. Circ Res. 1955 Nov;3(6):623-32. doi: 10.1161/01.res.3.6.623. No abstract available. PMID 13270378
- [Derived] Hassan AKM, Shaamash AH, Mohamed AG, Demitry SR, Razik NA. Comparison between invasive and non-invasive assessment of blood pressure in hypertensive disorders of pregnancy. Egypt Heart J. 2021 May 25;73(1):48. doi: 10.1186/s43044-021-00172-7. PMID 34032932